CLINICAL TRIAL: NCT06252116
Title: Study of Analgesic Action of Pregabalin, Duloxetine and Tramadol in Patients With Different Neuropathic Pain Phenotypes. Clinical Study
Brief Title: Study of Analgesic Action of Pregabalin, Duloxetine and Tramadol in Patients With Different Neuropathic Pain Phenotypes
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: 3/28
Record Dates: First submitted 2024-01-21; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuropathic pain patients: Patients were randomized to pregabalin (group A) and duloxetine (group B). Those patients who did not have a 50% reduction in pain levels received duloxetine (group A) and pregabalin (group B). Then, those patients who did not have a 50% reduction in pain levels received tramadol.
  Interventions: Drug: Pregabalin group; Drug: Duloxetine group

INTERVENTIONS:
Drug: Pregabalin group — Pregabalin group
Drug: Duloxetine group — Duloxetine group

SUMMARY:
Chronic pain is the most frequent cause from which millions of patients suffer worldwide, which makes them unable to work but also greatly affects their quality of life. Chronic pain is a condition in itself. Neuropathic pain is a consequence of damage or disease of the peripheral or central nervous system and presents a heterogeneous clinical profile. A large number of pharmaceutical and non-pharmacological agents, as well as various complementary therapies, have been used in the treatment of neuropathic pain. However, their effectiveness is considered moderate and limited and is under investigation because a significant proportion of patients do not respond satisfactorily to treatment.

Purpose: The purpose of the study is to investigate the effectiveness of analgesics in the different phenotypes of neuropathic pain.

DETAILED DESCRIPTION:
The existence of somatosensory nervous system damage and the consequent occurrence of neuropathic pain is an important factor in the development of many painful syndromes, both benign and cancerous pain. A particular feature of this syndrome is that patients with the same pathology (eg painful diabetic neuropathy) exhibit a different spectrum of symptoms and clinical signs whereas patients with different pathologies (such as diabetic neuropathy and postherpetic neuralgia) often have the same clinical picture. This phenomenon has been attributed to the different pathophysiological mechanisms involved in each case, regardless of the initial causative agent that induced the nerve damage. Among these mechanisms the occurrence of ectopic electrical activity in the periphery, the development of central sensitization, spinal cord remodeling as well as the phenotypic differentiation of neurons are included. In the treatment of neuropathic pain, a large number of agents have been used, such as antiepileptics, antidepressants, topical anesthetics, opioids, capsaicin etc. Among these, the highest efficacy, based on existing evidence, is proved with gabapentinoids (Gabapentin and Pregabalin) and antidepressants (serotonin and noradrenaline reuptake inhibitors) as well as Tramadol. The distinction of different phenotypes of neuropathic pain is done either by using specific questionnaires or by laboratory assessment. Regarding the use of questionnaires, the PAIN DETECT questionnaire has been used to distinguish 5 different phenotypes of neuropathic pain in patients with diabetic neuropathy, postherpetic neuralgia and back pain, and is considered as an acceptable method despite its limitations in the detection of different phenotypes of neuropathic painStudy protocol

Patients meeting the inclusion criteria are informed for and included in the study after written consent. Patients should note that this is an observational study and that the treatment they will receive is appropriate for their case, as documented in international guidelines. None will not receive an experimental or other medicine other than the medically accepted ones in their case and their treatment will be the same whether they are participating in the study or not. An initial assessment will be made to patients. During the initial assessment, demographic data, pain intensity with Numerical rating scale (NRS) and Short Form McGill Pain questionnaire, as well as location, reflections and periodicity are recorded. Additionally, patients are assessed on the basis of SOPA SF and PAIN Catastrophising scale questionnaires. Patients are then assessed for neuropathic pain with the DN4 and PAIN DETECT questionnaires. Since the latter are diagnostic of neuropathic pain, patients are divided into 2 groups. Group A begins to administer Pregabalin 50 mg daily with a gradual increase of 50 mg every 5 days to a dose of 300 mg daily or the highest tolerated dose based on adverse reactions. In group B, Duloxetin is administered at a dose of 30 mg, increasing to 60 mg daily after 15 days, in the absence of adverse events. Patients are re-evaluated after a 30-day NRS, McGill Pain questionnaire and PAIN DETECT scale for the range of sensory symptoms and signs. Since the reduction in pain intensity is less than 50% in the NRS, the second therapeutic agent is added as follows: Group A addition of Duloxetine at a dose of 30 mg, increasing to 60 mg daily after 15 days, in the absence of adverse effects. Group: Add Pregabalin 50mg with a gradual increase of 50mg per 5 days to a daily dose of 300mg or up to the maximum tolerated dose. Patients are re-evaluated 30 days after the addition of the second agent based on the NRS scale, McGill Pain Questionnaire and PAIN DETECT on the range of sensory symptoms and signs. Since the reduction in pain intensity is less than 50% in the NRS, the combination of the two agents in the two groups is added Tramadol 50 mg twice a day. Patients are re-evaluated after the latency of one month after the addition of Tramadol, and the final values in the NRS, PAIN DETECT SF McGill ranges are obtained. If at any stage of the treatment one of the drugs is not tolerated, it is discontinued, the patients are withdrawn from the study and by further measurements the case is recorded and the patient's alternative treatment methods are discussed with the patient.

Ethics

The study is a prospective cohort-type observational study and will include the recording of patients' clinical parameters without affecting their health, influencing the diagnostic or therapeutic approach, affecting the outcome of their health or violating their legal rights. Patient data will be recorded anonymously, and any publication of the results will take place in the form of aggregated tables, which does not contradict the personal or religious beliefs of patients.

ELIGIBILITY:
Inclusion Criteria:

* neuropathic pain

Exclusion Criteria:

* under 18 years old
* cancer pain
* patients receiving pregabalin, duloxetine, tramadol
* drug or alcohol abuse
* psychiatric decease
* renal failure, heart failure, liver failure, thrombocytopenia, closed-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from neuropathic pain (initial assessment with DN4 questionnaire)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
NRS Scale assessment | 1 month
  The initial assessment of the patients will be performed with the Numeric Rating Scale (NRS scale). NRS pain scale is a measure of pain intensity, in which the respondent selects a number from 0-10 that best reflects the intensity of his/her pain.

SECONDARY OUTCOMES:
Phenotype assessment | 1 month
  Pregabalin, duloxetine and tramadol that are prescribed for patients suffering from neuropathic pain affect different phenotypes of neuropathic pain regardless of the initial cause of pain. In this study we will examine and measure the affect of these agents on different symptoms of neuropathic pain burning sensation, tingling or prickling, pain touching, electric shock attacks, painful cold or heat water, numbness sensation, slight pressure pain. (scale from "NEVER" to "VERY STRONGLY".

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterini Amaniti, MD, PhD, Study Director — AHEPA University Hospital of Thessaloniki, Greece
Locations (1):
- AHEPA University General of Thessaloniki, Chronic Pain Unit, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campbell JN, Meyer RA. Mechanisms of neuropathic pain. Neuron. 2006 Oct 5;52(1):77-92. doi: 10.1016/j.neuron.2006.09.021. PMID 17015228
- [Background] Freeman R, Baron R, Bouhassira D, Cabrera J, Emir B. Sensory profiles of patients with neuropathic pain based on the neuropathic pain symptoms and signs. Pain. 2014 Feb;155(2):367-376. doi: 10.1016/j.pain.2013.10.023. Epub 2013 Oct 25. PMID 24472518
- See also: Peripheral neuropathic pain: from mechanisms to symptoms — https://pubmed.ncbi.nlm.nih.gov/10870735/
- See also: Usefulness and limitations of quantitative sensory testing: clinical and research application in neuropathic pain states — https://pubmed.ncbi.nlm.nih.gov/17451879/